CLINICAL TRIAL: NCT00131456
Title: Marijuana Addiction and Depression: Venlafaxine Treatment
Brief Title: Free Venlafaxine Treatment for Marijuana Addiction and Depression - 1
Acronym: VEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #4695; R01DA015451 (NIH)
Record Dates: First submitted 2005-08-16; First posted 2005-08-18 (Estimated); Results first posted 2013-06-04 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Depression; Marijuana Abuse
Keywords: cannabis dependence; depression; treatment; venlafaxine
MeSH Terms: conditions — Depression; Marijuana Abuse | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Venlafaxine (Active Comparator): Venlafaxine
  Interventions: Drug: Venlafaxine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Venlafaxine — 375mg/day
  Other Names: Effexor
  Arms: Venlafaxine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if Venlafaxine Extended Release (Ven-XR) is effective in treating individuals with marijuana addiction and depression.

DETAILED DESCRIPTION:
Given that depression and marijuana addiction often occur together, medications to treat individuals diagnosed with both conditions may be effective. The purpose of this study is to determine the effectiveness of Ven-XR in treating individuals diagnosed with depression and marijuana addiction.

During this twelve-week, double-blind, placebo-controlled study, study visits will occur twice each week. During study visits, participants will receive either placebo or medication and provide a urine sample for drug screening. Blood tests will be collected each month and women must take pregnancy tests each month. Throughout the study, all participants will receive individualized psychotherapy sessions. At each study visit, participants will be given $5 to cover transportation costs.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for current marijuana addiction and reports marijuana as primary drug of abuse
* Currently meets criteria for major depression or dysthymic disorder and receive a score of greater than or equal to 12 on the Hamilton Depression Inventory
* Clinically depressed for at least 3 months during a period of active marijuana use
* Women of child-bearing age will be included provided that they are not pregnant, based on the results of a blood pregnancy done at the time of screening and agree to use a method of contraception with proven efficacy and not to become pregnant during the study. To confirm this, blood pregnancy tests will be repeated monthly. Women will be provided a full explanation of the potential dangers of pregnancy while on the study. If a woman becomes pregnant, the study medication will be discontinued.

Exclusion Criteria:

* Meets criteria for past manic or psychotic disorder, unless substance-related
* History of a seizure disorder
* Individuals with chronic organic mental syndrome
* Any significant risk for suicide based on current assessment and history of attempts
* History of allergic reaction to either Venlafaxine or Ven-XR
* Unstable physical disorders that might make participation hazardous, such as uncontrolled hypertension and tachycardia (SBP>150, DBP >90, or a sitting quietly HR>100), acute hepatitis (patients with chronic mildly elevated transaminase levels (<2x upper limit of normal are acceptable) or unstable diabetes
* History of failure to respond to a previous adequate trial of Venlafaxine of at least 300 mg. for at least a 6-week period
* Physical dependence on any other drugs (excluding nicotine) that would require medical detoxification
* Currently being prescribed psychotropic medication by another physician (in the last 3 weeks), except for acute treatment of insomnia.
* Pregnant or breast-feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2004-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Levin, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: Click here for the Substance Treatment and Research Service website — http://www.stars.columbia.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from January 2004 through September 2010. Treatment seekers for problems related to marijuana use were recruited by local advertising or clinical referrals. Participants were treated at Columbia University/New York State Psychiatric Institute or at Columbia University/North Shore-LIJ Medical Center.
Pre-assignment Details: The trial included a one-week placebo lead-in. Placebo responders during the placebo lead in (N = 7), defined as a Clinical Global Impression rating of 1 or 2 and a reduction in the Hamilton Depression score > 75% or total score ≤ 7, were not randomized. Additionally, 13 participants were lost to follow-up so a total of 103 were randomized.
Groups:
- Placebo: Matched Placebo
- Venlafaxine: Venlafaxine: VEN-XR was titrated to the target dose of 225 mg/day (or the maximum tolerated dose) over the three weeks after randomization. After the fourth week post-randomization, patients with persistent depression who were not rated as having a CGI-Depression score of 1 ("very much improved') and who were tolerating 225 mg/day had their dose increased to a maximum of 375 mg/day.
Period: Overall Study
Arm/Group | Placebo | Venlafaxine
Started | 52 | 51
Completed | 33 | 31
Not Completed | 19 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Venlafaxine | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 51 | 103
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (9.3) | 34.2 (10.8) | 35.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 41 | 35 | 76
Region of Enrollment [Number; unit: participants]
  United States | 52 | 51 | 103

OUTCOME MEASURES:

1. Primary Outcome: Two Consecutive Weeks of Marijuana Abstinence
Description: The primary outcome measure for marijuana use was a dichotomous abstinence response,defined as at least two consecutive urine-confirmed abstinent weeks. Each week during the study, subjects were scored as urine-confirmed abstinent if both self-reported marijuana use for that week was negative, according to the quantitative substance use daily inventory (Timeline FollowBack), and all urines collected for that week were negative for THC. Patients who achieved the two consecutive abstinent weeks were classified as abstinent whether or not they subsequently dropped out of the study. Patients who dropped out of the study without achieving two continuous weeks of abstinence were classified as not abstinent.
Time Frame: measured daily by self report for 12 weeks of the trial or length of study participation
Population: All analyses were conducted based on the intent-to-treat principle.
Measure: Number; unit: participants
Arm/Group | Placebo | Venlafaxine
Number analyzed (Participants) | 52 | 51
participants | 19 | 6
Statistical Analysis 1: Comparison: Placebo vs Venlafaxine; Logistic regression was used to analyze all dichotomous outcomes. The dichotomous primary outcome marijuana abstinence was modeled using independent predictors: treatment(Venlafaxine vs. Placebo) and baseline urine THC level. The initial analysis included an interaction between treatment and baseline urine THC levels which was deemed not significant and omitted from the final logistic model; Test type: Superiority or Other; p < 0.01, Regression, Logistic

ADVERSE EVENTS:
Arm/Group | Placebo | Venlafaxine
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 24/52 | 33/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=52) | Venlafaxine (N=51)
anxiety (Psychiatric disorders) | 1 (1) | 6 (6)
diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (4)
dizziness (General disorders) | 2 (2) | 8 (8)
fatigue (General disorders) | 1 (1) | 6 (6)
GI Upset (Gastrointestinal disorders) | 2 (2) | 6 (6)
headache (General disorders) | 4 (4) | 2 (2)
insomnia (General disorders) | 4 (4) | 7 (7)
loss of libido (General disorders) | 0 (0) | 6 (6)
muscle aches (General disorders) | 4 (4) | 2 (2)
nausea (Gastrointestinal disorders) | 4 (4) | 6 (6)
syncopy or light headedness (General disorders) | 4 (4) | 2 (2)

LIMITATIONS AND CAVEATS:
This was an outpatient study and excluded patients with very severe depression. Thus we cannot generalize the findings to individuals with more severe depressive symptoms. The study length was relatively brief.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes